CLINICAL TRIAL: NCT02381990
Title: Office Based MRI/Ultrasound Guided Prostate Cryotherapy: Outcomes Registry
Brief Title: MRI/Ultrasound Fusion Guided Prostate Cryotherapy
Acronym: FIPC
Status: Recruiting | Type: Observational
Sponsor: Urological Research Network, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: URN-13-1010
Record Dates: First submitted 2015-01-12; First posted 2015-03-06 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Neoplasms Prostate; Cancer of the Prostate
Keywords: Prostate; PSA; FUSION; Ultrasound; MRI; Cancer; Cryotherapy; Outcomes; Recurrence; QOL, Quality of Life; Urinary function; Sexual Function
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: FUSE IMAGE MRI GUIDED PROSTATE CRYOTHERAPY — Biopsy proven Prostate Cancer is delimited and defined by MP-MRI. The MRI study is fused with transrectal ultrasound in realtime. The cryogenic "cryoprobes/devices" are employed to freeze and all "circuled or noted" cancer lesions. Two freeze 8 min/ thaw 10 min clycles are performed. Thermocouples are used to monitor treatment areas and safety margins
  Other Names: Intervention of Interest: Prostate Cryoablation

SUMMARY:
Registration of Prostate Cancer patients undergoing Prostate Cryotherapy guided by Mutiparametric-MRI (MP-MRI) highlighting biopsy confirmed regions. The primary outcome measure is 5 year oncological control. Secondary aim is lack of progression beyond the prostate gland. The aim of intervention is to eradicate prostate cancer disease in the treated area while imposing no or minimal deleterious effects in quality of life.

DETAILED DESCRIPTION:
CLINICAL TRIAL OF OBSERVATION NATURE

PRIMARY OUTCOME

Cancer control of treated areas 5, 10, 15 years after intervention based on prostate biopsy of initial treated area, progression requiring conversion to radical prostate surgery or radiation or other forms of whole gland treatment (ej, HIFU), Metastatic Free survival: CT Scan and Bone Scans, Cancer-Specific and Overall Survival

SECONDARY OUTCOMES

Secondary Interventions focal interventions due to de-novo lesions. Focal or target therapy rescue with other technologies (ej HIFU); Short, Intermediate and Long-Term Urinary and Sexual Function changes in quality of life measured by validated inventories; Anxiety related to cancer and cancer control. Treatment tolerance to local anesthesia. Patient App compliance and activity to monitor care

DATA COLLECTION

* Complete H&P, family history, past medical and surgical history, social history, allergies, and medications
* As of July 2016, voluntary measurement thru Focalyx App for smartphones and tablets
* Imaging Specifics Assessing Prostate, Seminal Vesicles and Urethral Contouring by Multi-parametric-MRI. Dominant lesions and secondary lesions contouring my MP-MRI.
* Procedure specific Co-Registration quality with ultrasound denoting quality
* Specific ablative description and digitalization of critical measures such as: ablation type (ej cryotherapy, equipment used) procedure, cryoprobes used, freeze/thaw cycles timing, temperatures at neurovascular bundles, denonvilliers fascia. Urethral warmer requirements
* Follow up information: 30 day perioperative outcomes (incidence of UTI, urinary retention, failure of local anesthetic, pain measures). 6 week, 3,6,9,12 month and then every 6 month measures of PSA, Testosterone levels, Urinary Function and Sexual Function inventories, Overall anxiety and regret related to diagnosis and treatment
* Uroflow and PVR measurements by 3 to 6 month of treatment
* MP MRI on a yearly basis, for years 2,3,4 after treatment, biopsy driven by new suspicious MRI findings
* MP MRI triggered by elevation in PSA velocity or PSA level 10% above diagnosis
* Transperineal Fusion Guided Prostate biopsy at 1st year - emphasis on treated areas, suspicious MRI areas
* Transperineal Fusion Guided Prostate biopsy at 5th year - emphasis on treated areas, suspicious MRI areas
* 5, 10, 15 Yr CT Scans, PET Scan/Bone Scan

SAFETY MEASURES

* Periodic evaluation of registry to ensure consistency in follow up
* Patient remainders of tests required

ELIGIBILITY:
Inclusion Criteria:

* Men between 55 and 65 years of age with a clinical diagnosis of prostate cancer with Low or Intermediate risk prostate cancer, and <50% positive core rate by prostate lobe
* Men older than 65 years of age with clinical diagnosis of prostate cancer <50% positive core rate by prostate lobe
* Absence of extra-capsular extension
* Absence of seminal vesicle invasion
* Absence of regional or distant metastatic disease
* Multiparametric MRI of the prostate performed either before the biopsy or >10 weeks after prostate biopsy
* Treated with Cryotherapy of the prostate
* Treatment based on co-registration between MP-MRI and Prostate Ultrasound

Exclusion Criteria:

* Prior treatment of prostate cancer in the form of surgery.
* Performance status greater than 0 based on ECOG criteria
* Mental status impairment

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As written in Initial Section
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2033-08 (Estimated)

PRIMARY OUTCOMES:
Oncological Control | 1 Year
  Lack of prostate cancer presence in treated area after MRI/US FUSION Biopsy

SECONDARY OUTCOMES:
Oncological Control | 1 Year
  Lack of prostate cancer presence in the gland after MRI/US FUSION Biopsy
Oncological Control | Yearly, up to 10 years
  Lack of prostate cancer presence in gland measured by MP-MRI
Urinary Functional Outcomes | Every 3 months up to 24 months
  Evaluation of urinary function outcomes when compared to baseline using expanded prostate composite index and AUA symptoms scores. Urinary function also by objective measurements - uroflow and post void residuals
Perioperative Outcomes | 30 days
  Procedure tolerance, need for hospital admission or ER consultation, incidence of urinary tract infection, urinary retention, any significant side effect that may occur and perioperative survivel
Sexual Functional Outcomes | Every 3 months up to 24 months
  Evaluation of sexual function outcomes when compared to baseline using Sexual Inventory for men questionnaires

OTHER OUTCOMES:
Secondary Treatment Requirement | Yearly, up to 10 years
  Type of treatments required after initial intervention over time

CONTACTS AND LOCATIONS:
Overall Officials: FERNANDO J BIANCO, MD, Principal Investigator — UROLOGICAL RESEARCH NETWORK; EUSEBIO LUNA, MD, Study Director — UROLOGICAL RESEARCH NETWORK; Isabel H Lopez, MD, Study Director — UROLOGICAL RESEARCH NETWORK
Locations (1):
- Urological Research Network, Miami Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Non identifiable pertinent information will be shared for other scientists to evaluate other pertinent questions

REFERENCES:
- [Result] Moore CM, Kasivisvanathan V, Eggener S, Emberton M, Futterer JJ, Gill IS, Grubb Iii RL, Hadaschik B, Klotz L, Margolis DJ, Marks LS, Melamed J, Oto A, Palmer SL, Pinto P, Puech P, Punwani S, Rosenkrantz AB, Schoots IG, Simon R, Taneja SS, Turkbey B, Ukimura O, van der Meulen J, Villers A, Watanabe Y; START Consortium. Standards of reporting for MRI-targeted biopsy studies (START) of the prostate: recommendations from an International Working Group. Eur Urol. 2013 Oct;64(4):544-52. doi: 10.1016/j.eururo.2013.03.030. Epub 2013 Mar 20. PMID 23537686
- [Result] Bahn D, de Castro Abreu AL, Gill IS, Hung AJ, Silverman P, Gross ME, Lieskovsky G, Ukimura O. Focal cryotherapy for clinically unilateral, low-intermediate risk prostate cancer in 73 men with a median follow-up of 3.7 years. Eur Urol. 2012 Jul;62(1):55-63. doi: 10.1016/j.eururo.2012.03.006. Epub 2012 Mar 21. PMID 22445223
- [Result] Costa DN, Pedrosa I, Donato F Jr, Roehrborn CG, Rofsky NM. MR Imaging-Transrectal US Fusion for Targeted Prostate Biopsies: Implications for Diagnosis and Clinical Management. Radiographics. 2015 May-Jun;35(3):696-708. doi: 10.1148/rg.2015140058. Epub 2015 Mar 18. PMID 25786055
- [Result] Barentsz JO, Richenberg J, Clements R, Choyke P, Verma S, Villeirs G, Rouviere O, Logager V, Futterer JJ; European Society of Urogenital Radiology. ESUR prostate MR guidelines 2012. Eur Radiol. 2012 Apr;22(4):746-57. doi: 10.1007/s00330-011-2377-y. Epub 2012 Feb 10. PMID 22322308
- [Result] Siddiqui MM, Rais-Bahrami S, Turkbey B, George AK, Rothwax J, Shakir N, Okoro C, Raskolnikov D, Parnes HL, Linehan WM, Merino MJ, Simon RM, Choyke PL, Wood BJ, Pinto PA. Comparison of MR/ultrasound fusion-guided biopsy with ultrasound-guided biopsy for the diagnosis of prostate cancer. JAMA. 2015 Jan 27;313(4):390-7. doi: 10.1001/jama.2014.17942. PMID 25626035